CLINICAL TRIAL: NCT00803855
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Single Ascending Dose Study to Asses the Safety, Tolerability, Pharmacokinetics of AZD1446 Including an Open Food Effect Panel in Healthy Male and Non-Fertile Female Volunteers
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics After Single Doses of AZD1446 to Healthy Volunteers
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Didier Meulien, MD, PhD, Medical Science Director, Clinical Neuroscience, Therapeutic area Alzheimers Disease and Cognition, AstraZeneca R&D Södertälje
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: D1950C00001; EudraCT No.: 2008-006228-76
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: single dose; pharmacokinetics; safety; healthy volunteers; food interaction; AZD1446
MeSH Terms: interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1446 Oral or placebo (Experimental): Single oral administration of AZD1446 or placebo
  Interventions: Drug: AZD1446
- AZD1446 Oral, with or without food (Experimental): Single oral administration of AZD1446 with or without food
  Interventions: Drug: AZD1446

INTERVENTIONS:
Drug: AZD1446 — oral, single dose

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of AZD1446 following single dose administration.

ELIGIBILITY:
Inclusion Criteria:

* physical healthy volunteers
* weight between 50 to 100 kg and a body mass index (BMI) between 19 and 30 kg/m2

Exclusion Criteria:

* History of any clinically significant disease or disorder.
* History of severe allergy/hypersensitivity reactions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD1446 by assessment of serious adverse events, ECGs, vital signs and laboratory variables | From first to last visit

SECONDARY OUTCOMES:
Determine the single ascending dose pharmacokinetics of AZD1446 | PK sampling taken at defined timepoints during residential period
Determine the single dose of AZD1446 on food interaction | From first to last visit

CONTACTS AND LOCATIONS:
Overall Officials: Didier Meulien, MD, PhD, MSD, Study Director — AstraZeneca Södertälje; Ingemar Bylesjö, MD, PhD, Principal Investigator — AstraZeneca CPU Huddinge
Locations (1):
- Research site, Huddinge, Sweden